CLINICAL TRIAL: NCT03927833
Title: Cycled Phototherapy: A Safer Effective Method to Control the Serum Bilirubin Of Extremely Premature Infants?
Brief Title: Cycled Phototherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NICHD-NRN-0061; UG1HD034216 (NIH); UG1HD027904 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD027851 (NIH); UG1HD087229 (NIH); UG1HD053109 (NIH); UG1HD068278 (NIH); UG1HD068244 (NIH); UG1HD068263 (NIH); UG1HD027880 (NIH); UG1HD053089 (NIH); UG1HD087226 (NIH); UG1HD112079 (NIH); UG1HD112097 (NIH); UG1HD112100 (NIH); 3U24HD095254-07 (NIH)
Record Dates: First submitted 2019-04-18; First posted 2019-04-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hyper Bilirubinemia; Premature Infant
Keywords: Infant, Newborn, Diseases; Phototherapy
MeSH Terms: conditions — Premature Birth; Infant, Newborn, Diseases

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized clinical trial addressing patient safety.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Phototherapy (Active Comparator): Continuous phototherapy
  Interventions: Device: Phototherapy lights
- Cycled Phototherapy (Experimental): Cycled phototherapy at timed intervals, dependent upon total serum bilirum (TSB) levels.
  Interventions: Device: Phototherapy lights

INTERVENTIONS:
Device: Phototherapy lights — Phototherapy lights used continuously or timed, following an algorithm based upon TSB levels.

SUMMARY:
Cycled phototherapy (PT) is likely to increase survival over that with continuous PT among extremely premature infants (< 750 g BW or <27 weeks GA).

DETAILED DESCRIPTION:
Were they not delivered early, extremely premature infants would normally develop in darkness within the uterus for 3-4 more months longer before birth. Yet, the routine care of these infants has involved the use of uninterrupted (continuous) exposure to bright light during phototherapy (PT), a treatment method that neonatologists have assumed has no serious adverse effects on even the most immature of newborns.

Immaturity, thin translucent skin, and a multitude of other problems may make extremely premature infants highly vulnerable to the photo-oxidative injury, lipid peroxidation, DNA damage, reduced cerebral and mesenteric blood flow, or other serious potential hazards of uninterrupted exposure to PT that have now been identified. Such hazards were not recognized when continuous PT was widely incorporated into neonatal care, and the survival rate of extremely premature infants (<27 wks gestation or <750 g birth weight) was much lower than today.

PT rapidly photoisomerizes bilirubin in the subcutaneous tissues and vasculature, and six trials of cycled PT have demonstrated that use of cycled PT reduces the total hours of PT and results in minimal or no increase in peak TSB over that with continuous PT in term or moderately preterm infants. Recent findings from a pilot study (NCT01944696) support a PT regimen for this Cycled Phototherapy protocol.

Infants born at one of the Neonatal Research Network centers, ≤ 750 grams at birth and/or < 27 weeks gestation at birth by best OB estimate will be considered for this study.

Those who qualify will be randomized to either cycled PT or continuous PT. The cycled phototherapy begins with >15 min/h cycled PT regimen and increased to 30 min/h if the TSB is 8.0-9.9 and 60 min/h if the TSB is >10 mg/dL. Those randomized to continuous phototherapy will undergo continuous exposure,as that is commonly used in NRN centers.

The PT lamp position will be adjusted to meet the irradiance (µW/cm2/nm) goal of 22 at the umbilicus. The irradiance goal in both groups will be increased from 22 to 33 at a TSB of 10-13 and to 40 at a TSB >13.

ELIGIBILITY:
Inclusion Criteria:

1. Infants is inborn
2. Infant is ≤ 750 grams at birth and/or < 27 weeks gestation at birth by best OB estimate
3. Infant is 12-36 hours of age.

Exclusion Criteria:

1. Unable to enroll infant by 36 hours of age
2. Previous phototherapy
3. Known hemolytic disease
4. TSB reported as >6.0 mg/dL before 12 hours age
5. Major anomaly
6. Overt nonbacterial infection
7. Infant is likely to expire soon: Limiting or withdrawal of intensive care is being recommended to the parents, the parents are requesting withdrawal of care, or the pH is < 6.80 or persistent bradycardia with hypoxemia for >2h.

Ages: 22 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1700 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants survival to discharge | Birth to hospital discharge, up to 120 days of life
  Number of Participants discharged from hospital alive, after birth.

SECONDARY OUTCOMES:
Number of hours of Phototherapy | Start until the end of intervention period (duration of 2 weeks)
  The reported values will be the mean total hours of phototherapy during the two week intervention period.
Number of irradiance hours | Start until the end of intervention period (duration of 2 weeks)
  The reported values will be the mean total hours of irradiance during the two week intervention period.
Peak Concentration of Total Serum Bilirubin | Start until the end of intervention period (duration of 2 weeks)
  The reported values will be the mean peak total serum bilirubin (mg/dL) during the two week intervention period.
Concentration of Total Serum Bilirubin | Start until the end of intervention period (duration of 2 weeks)
  The reported values will be the mean total serum bilirubin (mg/dL) during the two week intervention period.
Number of Participants with Major neonatal morbidity | Birth to hospital discharge, up to 120 days of life
  Major neonatal morbidity is defined as a severe ICH, ventricular enlargement of cystic white matter disease, BPD, late onset sepsis, NEC or spontaneous intestinal perforation, or >grade 3 ROP before discharge.
Number of Participants with Severe ICH, as a component of the predischarge morbidity | Birth to hospital discharge, up to 120 days of life
  As recorded for the sonongram with the most severe finding in the blood/echodensity in the ventricle or blood/echodensity in the parenchyma
Number of Participants with Ventricular enlargement of cystic white matter disease, as a component predischarge morbidity | Birth to hospital discharge, up to 120 days of life
  If a MRI was done: ventricular size enlarged, cystic PVL or porencephalic /posthemorrhagic cyst/multicystic encephalomalacia observed. If a MRI was not done: the same items as above for sonograms after day 28.
Number of Participants with Bronchopulmonary dysplasia (BPD), as a component predischarge morbidity | Birth to hospital discharge, up to 120 days of life
  BPD defined as highest FiO2 at 36 wk: >0.21
Number of Participants with Late onset sepsis, as a component predischarge morbidity | Birth to hospital discharge, up to 120 days of life
  Late onset blood culture positive septicemia/bacteremia at >72 hours of age.
Number of Participants with Necrotising enterocolitis (NEC) or spontaneous intestinal perforation, as a component predischarge morbidity | Birth to hospital discharge, up to 120 days of life
  Either proven NEC or spontaneous gastrointestinal perforation without proven NEC.
Number of Participants with Grade 3 (or greater) retinopathy of prematurity (ROP), as a component predischarge morbidity | Birth to hospital discharge, up to 120 days of life
  Stage 3 ROP observed in either eye.
Number of Participants with Patent ductus arteriosus (PDA) treated with surgery or NSAIDS | Birth to hospital discharge, up to 120 days of life
  PDA treated with surgery or NSAIDS (indomethacin, ibuprofen or acetaminophen)
Number of Participants with Neurodevelopmental Impairment | Birth to 26 months corrected age
  Neurodevelopmental Impairment (NDI), as assessed in a sub-population of follow-up of infants <27 wks gestation. Severe NDI will be defined by any of the following: a BSID III cognitive score < 70, Gross Motor Functional (GMF) Level of 3-5, blindness (<20/200 vision) or profound hearing loss (inability to understand commands despite amplification); moderate NDI will be defined as a BSID III cognitive score 70-84 and either a GMF level of 2 or a hearing deficit requiring amplification to understand commands or unilateral blindness; mild NDI will be defined by a cognitive score 70-84, or a cognitive score ≥ 85 and any of the following: presence of a GMF level 1 or hearing loss not requiring amplification. Normal (no NDI) will be defined by a cognitive score ≥ 85 and absence of any neurosensory deficits.
Number of Participants with Neurodevelopmental Impairment or Death | Birth to 26 months corrected age
  NDI defined in outcome #9

CONTACTS AND LOCATIONS:
Overall Officials: Jon Tyson, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Mississippi Medical Center - Children's of Mississippi, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov)